CLINICAL TRIAL: NCT07315269
Title: Evaluation of the Effect of Daytime Power Napping on Depression, Stress and Sleep According to Working Method: Prospective Cohort Study
Brief Title: The Relationship Between Power Sleep and Sleep Quality, Depression, and Stress Levels in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: okkes zortuk (Other)
Responsible Party: Sponsor-Investigator, okkes zortuk, Manager, Ataturk University
Organization: Ataturk University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZTKLAB003102022DSEC23092022237
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2023-12

CONDITIONS: Sleep Quality; Depression Disorders; Stress, Psychological; Occupational Stress
Keywords: Naps; Power napping; Shift workers; Daytime sleep; Mental health; Prospective cohort study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress, Psychological; Occupational Stress; Psychological Well-Being

STUDY DESIGN:
Masking Description: Daytime Power Nap Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daytime Power Nap Group (Experimental): A group of 40 participants who are instructed to perform a 15-20 minute power nap daily for 6 weeks.
  Interventions: Behavioral: Daytime Power Napping

INTERVENTIONS:
Behavioral: Daytime Power Napping — The duration, effectiveness, and method of intervention in this area should be clearly stated:
  Duration Per Session: Each nap is planned to be between 15-20 minutes, and limited to a maximum of 30 minutes to prevent sleepiness (sleep inertia).
  Total Duration: The intervention is a 6-week process. Target Group: 40 healthy volunteers (including day and shift workers). Goal: To enhance the privacy of sleep in daily life, reduce virus spread, and decrease stress.

SUMMARY:
This prospective cohort study aims to evaluate the effects of daily daytime power napping on sleep quality, depression, and perceived stress levels among healthy individuals. The study particularly investigates whether these effects differ between daytime workers and shift workers. Participants are required to practice a 15-20 minute (maximum 30 minutes) power nap daily for a period of six weeks. Changes in psychological and sleep parameters are assessed using the Jenkins Sleep Scale (JSS), Beck Depression Scale (BDS), and Perceived Stress Scale (PSS) before and after the intervention.

DETAILED DESCRIPTION:
The study was conducted with 40 healthy volunteers (including 29 daytime workers and 11 shift workers) to analyze the impact of daytime napping on mental health and sleep hygiene.

Methodology: At the beginning of the study, participants' demographic information was collected, and baseline assessments were performed using the Jenkins Sleep Scale (JSS) for sleep patterns, the Beck Depression Scale (BDS) for depressive symptoms, and the Perceived Stress Scale (PSS) for stress levels.

Intervention: Participants were instructed to take a short nap (power nap) between 1:00 PM and 3:00 PM for daytime workers, or at suitable intervals for shift workers, every day for 6 weeks. The duration of the nap was strictly limited to 15-30 minutes to avoid sleep inertia.

Evaluation: After the 6-week intervention period, the same scales (JSS, BDS, and PSS) were administered as a post-test. The data were analyzed to compare the pre-test and post-test scores, with a focus on the differences in outcomes between different work schedules (shift vs. daytime). The study adheres to the principles of the Declaration of Helsinki and was approved by the Dicle University Social Sciences and Humanities Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy volunteer.
* Being actively employed as either a daytime worker or a shift worker.
* Providing written informed consent to participate in the study.
* Willingness to adhere to a 6-week daytime power napping protocol.

Exclusion Criteria:

* Presence of diagnosed severe sleep disorders (e.g., severe insomnia or sleep apnea) that might interfere with the study protocol.
* Inability to complete the 6-week power napping intervention.
* Missing or incomplete psychological scale data at baseline or post-test.
* Failure to perform the power nap as instructed during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Quality as measured by the Jenkins Sleep Scale | Baseline (Day 0) and at the end of the 6-week intervention period.
  The JSS is a 4-item scale used to assess sleep problems, specifically focusing on difficulties falling asleep and maintaining sleep quality. Each item is scored on a 6-point Likert scale (0-20 total range). Higher scores indicate more sleep problems.

SECONDARY OUTCOMES:
Change in Depressive Symptoms as measured by the Beck Depression Scale (BDS/BDI) | Baseline (Day 0) and at the end of the 6-week intervention period.
  The BDS consists of 21 questions designed to assess cognitive, somatic, and emotional symptoms of depression. Scores range from 0 to 63. Higher scores indicate more severe depressive symptoms.
Change in Perceived Stress as measured by the Perceived Stress Scale (PSS). | Baseline (Day 0) and at the end of the 6-week intervention period.
  The 10-item version of the PSS measures an individual's perception of stress in their current situation. It includes two sub-dimensions: "perception of inadequate self-efficacy" and "perception of stress discomfort". Higher scores indicate a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ökkeş Zortuk, Principal Investigator — Emergency Medicine Department, Defne Government Hospital; Yeşim Dersuneli, MSc, Study Director — Clinical Psychology, Muş Alparslan University; Özlem Tolan, PHd, Study Chair — Clinical Psychology, Dicle University
Locations (1):
- Dicle University, Diyarbakır, Diyarbakar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To maintain participant confidentiality and comply with the institutional ethics committee's guidelines, individual participant data (IPD) will not be made publicly available. However, metadata and study results are reported within the manuscript.

REFERENCES:
- [Background] Brown JP, Martin D, Nagaria Z, Verceles AC, Jobe SL, Wickwire EM. Mental Health Consequences of Shift Work: An Updated Review. Curr Psychiatry Rep. 2020 Jan 18;22(2):7. doi: 10.1007/s11920-020-1131-z. PMID 31955278
- [Background] Faraut B, Boudjeltia KZ, Dyzma M, Rousseau A, David E, Stenuit P, Franck T, Van Antwerpen P, Vanhaeverbeek M, Kerkhofs M. Benefits of napping and an extended duration of recovery sleep on alertness and immune cells after acute sleep restriction. Brain Behav Immun. 2011 Jan;25(1):16-24. doi: 10.1016/j.bbi.2010.08.001. Epub 2010 Aug 8. PMID 20699115
- [Result] Juhola J, Arokoski JPA, Ervasti J, Kivimaki M, Vahtera J, Myllyntausta S, Saltychev M. Internal consistency and factor structure of Jenkins Sleep Scale: cross-sectional cohort study among 80 000 adults. BMJ Open. 2021 Jan 18;11(1):e043276. doi: 10.1136/bmjopen-2020-043276. PMID 33462100